CLINICAL TRIAL: NCT05622929
Title: A Pragmatic Cluster Randomized Trial to Assess the Effect of a Digitally Enabled Quality Improvement Intervention on LDL Cholesterol Control in Atherosclerotic Established Cardiovascular Disease Patients
Brief Title: Cluster Randomized Trial of a Digital Quality Improvement Intervention on LDLCholesterol Control
Acronym: SAPPHIRE-LDL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: epHealth primary care solutions (Unknown); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CKJX839A1BR05R; 63520022.6.1001.0071 (Other: CAAE)
Record Dates: First submitted 2022-11-14; First posted 2022-11-21 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-04

CONDITIONS: Cardiovascular Diseases; Atherosclerosis; Dyslipidemias
Keywords: Cardiovascular diseases; Atherosclerosis; Dyslipidemias
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis; Dyslipidemias

STUDY DESIGN:
Intervention Model Description: Cluster randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Real-world evidence (RWE) platform to provide data on their clinical practice + usual care + Digitally-enabled Multifaceted Quality Improvement Intervention
  Interventions: Behavioral: Digitally-enabled Multifaceted Quality Improvement Intervention
- Control group (Active Comparator): RWE platform to provide data on their clinical practice + usual care
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Digitally-enabled Multifaceted Quality Improvement Intervention — Digitally-enabled multifaceted strategy in addition to access to a RWE platform to provide clinical data. The digitally-enabled multifaceted strategy will include various tools that will provide support to the health professionals responsible for treating ASCVD patients in each center as well as patients, including:
  * Knowledge of effective lipid lowering therapies
  * Clinical decision support
  * Audit and feedback on adherence to optimal clinical management
  * Audit and feedback on LDL-C control
  Arms: Intervention group
Behavioral: Usual care — Health professionals responsible for treating ASCVD patients in each center will continue to provide usual care to ASCVD patients in addition to provide data through a RWE platform.
  Arms: Control group

SUMMARY:
Elevation in low density lipoprotein (LDL) cholesterol (LDL-C) is a causal risk factor for atherosclerotic established cardiovascular disease (ASCVD). Reduction of LDL-C with statins has been clearly demonstrated as a robust and cost-effective way of reducing the burden of ASCVD in individuals at risk. ASCVD is the leading cause of death and disability in Brazil and therefore prevention guidelines recommend LDL-C reduction with the aim of reducing disease burden in individuals at risk. Studies have shown a clear hiatus on awareness and treatment of cholesterol in Brazil. Thus, it became imperative to develop knowledge translation projects aiming at bridging the gap between science and clinical practice and ultimately leading to better outcomes. Cluster randomized clinical trials are the highest quality type of clinical research to test educational and active interventions aimed at changing behaviors or clinical practices. Therefore, this study is a pragmatic cluster randomized trial to assess the effect of a digitally enabled quality improvement intervention on LDL-C control in atherosclerotic established cardiovascular disease (ASCVD) patients.

DETAILED DESCRIPTION:
Elevation in low density lipoprotein (LDL) cholesterol (LDL-C) is a causal risk factor for atherosclerotic established cardiovascular disease (ASCVD). Reduction of LDL-C with statins has been clearly demonstrated as a robust and cost-effective way of reducing the burden of ASCVD in individuals at risk. ASCVD is the leading cause of death and disability in Brazil and therefore prevention guidelines recommend LDL-C reduction with the aim of reducing disease burden in individuals at risk. Studies have shown a clear hiatus on awareness and treatment of cholesterol in Brazil. Thus, it became imperative to develop knowledge translation projects aiming at bridging the gap between science and clinical practice and ultimately leading to better outcomes. Cluster randomized clinical trials are the highest quality type of clinical research to test educational and active interventions aimed at changing behaviors or clinical practices.To our knowledge, data from this study will be crucial to leverage LDL-C treatment in Brazil, considering efforts to improve population health. The present study represents one of the first trials testing a quality improvement (QI) intervention targeted to LDL-C reduction in ASCVD patients conducted in a middle-income country. These results will address whether the proposed QI intervention is feasible and effective in these settings. Therefore, this study is a pragmatic cluster randomized trial to assess the effect of a digitally enabled QI intervention on LDL-C control in ASCVD patients. This study will have 2 phases. Phase 1 will be an observational phase prior to randomization of clusters with the objective to assess the baseline LDL-C levels achieved for target patients. Phase 2 will be an interventional phase, in which clusters will be randomized to the digitally enabled quality improvement intervention or usual care, with the objective to assess the effect of a digitally enabled QI intervention on control of LDL-C levels in ASCVD patients.

ELIGIBILITY:
Patient Eligibility Criteria:

Inclusion Criteria:

* Capable of using a smartphone with iOS or Android System AND
* Established ASCVD, including:

  1. Coronary Artery Disease (CAD):

     * Prior myocardial infarction
     * Prior coronary revascularization - percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG)
     * Angiographic or computerized tomography (CT)-imaging evidence of coronary atherosclerosis (≥ 50% stenosis in at least one major epicardial coronary artery)
  2. Stroke:

     • Prior ischemic stroke thought not to be caused by an embolic cause (e.g., atrial fibrillation, valvular heart disease or mural thrombus)
  3. Peripheral Artery Disease (PAD):

     * Prior documentation of a resting ankle-brachial index ≤ 0.9
     * History of prior percutaneous or surgical revascularization of an iliac, femoral, or popliteal artery
     * Prior non-traumatic amputation of a lower extremity due to peripheral artery disease
     * History of prior percutaneous or surgical carotid artery revascularization
     * Carotid Stenosis > 50% on prior angiography or ultrasound AND
* Provision of informed consent

Exclusion Criteria:

* Patients with a recent cardiovascular event, less than 3 months prior to study inclusion
* Patients with LDL-C ≤ 50 mg/dL
* Current participation in other clinical trials involving lipid lowering treatments
* Patients that do not consent to trial participation

Cluster Eligibility Criteria:

Inclusion Criteria:

* Outpatient Clinics from public or private hospitals OR, Private Practices, which assist patients with previous ASCVD on secondary prevention that provide a unit/institution authorization form for participation in the trial AND
* Minimum monthly volume of 20 ASCVD patients

Exclusion Criteria:

* Clusters that do not provide the unit/institution authorization form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1465 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1: LDL-C levels | Baseline
  LDL-C levels measured at a single visit
Phase 2: LDL-C | 6 months
  LDL-C levels measured at the end of follow up of Phase 2

SECONDARY OUTCOMES:
Phase 1: Prescribed lipid-lowering therapy | Baseline
  Percentage of patients on prescribed lipid-lowering therapy
Phase 1: Prescribed combination lipid-lowering therapy | Baseline
  Percentage of patients on prescribed combination lipid-lowering therapy
Phase 1: Prescribed intensive lipid-lowering therapy | Baseline
  Percentage of patients on prescribed intensive lipid-lowering therapy
Phase 1: Prescription of any statins | Baseline
  Percentage of prescription of any statins
Phase 1: Prescription of high intensity statins | Baseline
  Percentage of prescription of high intensity statins
Phase 1: Prescription of ezetimibe | Baseline
  Percentage of prescription of ezetimibe
Phase 1: Prescription of PCSK9 monoclonal antibody or siRNA PCSK9 inhibitors | Baseline
  Percentage of prescription of PCSK9 monoclonal antibody or siRNA PCSK9 inhibitors
Phase 1: LDL-C < 50 mg/dL | Baseline
  Percentage of patients with LDL-C < 50 mg/dL
Phase 2: Prescribed lipid-lowering therapy | 6 months
  Percentage of patients on prescribed lipid-lowering therapy
Phase 2: Prescribed combination lipid-lowering therapy | 6 months
  Percentage of patients on prescribed combination lipid-lowering therapy
Phase 2: Prescribed intensive lipid-lowering therapy | 6 months
  Percentage of patients on prescribed intensive lipid-lowering therapy
Phase 2: Prescription of any statins | 6 months
  Percentage of prescription of any statins
Phase 2: Prescription of high intensity statins | 6 months
  Percentage of prescription of high intensity statins
Phase 2: Prescription of moderate intensity statins | 6 months
  Percentage of prescription of moderate intensity statins
Phase 2: Prescription of low intensity statins | 6 months
  Percentage of prescription of low intensity statins
Phase 2: Prescription of ezetimibe | 6 months
  Percentage of prescription of ezetimibe
Phase 2: Prescription of PCSK9 monoclonal antibody or siRNA PCSK9 inhibitors | 6 months
  Percentage of prescription of PCSK9 monoclonal antibody or siRNA PCSK9 inhibitors
Phase 2: LDL-C < 50 mg/dL | 6 months
  Percentage of patients with LDL-C < 50 mg/dL
Phase 2: LDL-C relative change | 6 months
  Change in LDL-C relative to baseline
Phase 2: LDL-C reduction of ≥50% | 6 months
  Percentage of patients with LDL-C reduction of ≥50% relative to baseline
Phase 2: non-HDL-C relative change | 6 months
  Change in non-HDL-C relative to baseline
Phase 2: Barriers for drug prescription | 6 months
  Barriers for drug prescription at the system (cluster) and physician level
Phase 2: Adherence to prescribed lipid-lowering therapy | 6 months
  Patient´s adherence to prescribed lipid-lowering therapy
Phase 2: Barriers for drug adherence | 6 months
  Patient´s barriers for drug adherence
Phase 2: Intolerance to Statins | 6 months
  Percentage of patients with intolerance to Statins

OTHER OUTCOMES:
Phase 2: 5P-MACE (Major Cardiovascular Events) | 6 months
  Composite endpoint of time to first occurrence of a major cardiovascular event 5P-MACE including cardiovascular deaths, non-fatal stroke or transient ischemic attack (TIA), non-fatal myocardial infarction, hospitalization for unstable angina, or coronary revascularization, whichever occurs first
Phase 2: 3P-MACE (Major Cardiovascular Events) | 6 months
  Composite endpoint of time to first occurrence of a major cardiovascular event 3P-MACE including cardiovascular deaths, non-fatal stroke or TIA, or non-fatal myocardial infarction, whichever occurs first
Phase 2: Cardiovascular death | 6 months
  Time to cardiovascular death
Phase 2: Death from any cause | 6 months
  Time to death from any cause
Phase 2: Myocardial infarction | 6 months
  Time to first myocardial infarction
Phase 2: Stroke | 6 months
  Time to first stroke
Phase 2: Coronary revascularization | 6 months
  Time to first coronary revascularization
Phase 2: Total deaths | 6 months
  Total deaths within 6 months from inclusion

CONTACTS AND LOCATIONS:
Overall Officials: M. Julia Machline-Carrion, PhD, Principal Investigator — epHealth
Locations (28):
- Brazil (28):
  - Hospital da Bahia, Salvador, Estado de Bahia
  - Hospital Santa Lúcia, Poços de Caldas, Minas Gerais
  - Hospital e Maternidade Angelina Caron, Campina Grande do Sul, Paraná
  - Hospital Regional Hans Dieter Schmidt, Joinville, Santa Catarina
  - Centro de Pesquisa Clínica do Coração, Aracaju, Sergipe
  - Hospital Universitário São Francisco de Assis, Bragança Paulista, São Paulo
  - Instituto de Pesquisa Clínica de Campinas, Campinas, São Paulo
  - Irmandade da Santa Casa de Misericórdia de Marilia, Marília, São Paulo
  - Hospital Carlos Fernando Malzoni, Matão, São Paulo
  - Hospital Universitário João de Barros Barreto, Belém
  - UPECLIN - Unidade de Pesquisa Clínica da Faculdade de Medicina de Botucatu, Botucatu
  - Santa Casa de Curitiba, Curitiba
  - Centro de Pesquisas em Diabetes e Doenças Endócrino-metabólicas, Fortaleza
  - Hospital Municipal de Aparecida de Goiânia, Goiânia
  - Hospital Ruy Azeredo, Goiânia
  - Centro de Pesquisas Clínicas Dr Marco Mota, Maceió
  - Instituto Atena de Pesquisa Clínica, Natal
  - Unidade Hospital Municipal Antônio Giglio, Osasco
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - Santa Casa de Porto Alegre, Porto Alegre
  - Hospital Regional Presidente Prudente, Presidente Prudente
  - Clínica Silvestre Santé, Rio Branco
  - Instituto Nacional de Cardiologia, Rio de Janeiro
  - Instituto de Cardiologia de Santa Catarina, São José
  - Hospital São Paulo (UNIFESP), São Paulo
  - Hospital São Paulo Universidade Federal de São Paulo, São Paulo
  - Instituto de Cardiologia Dante Pazzanese, São Paulo
  - Hospital Evangélico de Vila Velha, Vila Velha

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Machline-Carrion MJ, Girotto AN, Raupp P, Marton Pereira P, Monfardini F, Santos RD, Santo K, Ray K, Cannon CP, Berwanger O. Rationale, design and prerandomization data for a cluster randomized trial to assess the effect of a digitally enabled quality improvement intervention on LDL-C control in established atherosclerotic cardiovascular disease patients: The SAPPHIRE-LDL trial. Am Heart J. 2025 Jun;284:1-10. doi: 10.1016/j.ahj.2025.01.019. Epub 2025 Feb 3. PMID 39909341